CLINICAL TRIAL: NCT07258212
Title: Safety and Normative Data With Neos™, in Healthy Volunteers, Children and Patient Populations With Ophthalmological or Neurological Disease
Brief Title: Safety and Normative Data With Neos™
Acronym: neos-SNOW
Status: Recruiting | Type: Observational
Sponsor: machineMD AG (Industry)
Responsible Party: Sponsor
Other Study IDs: CI-001
Record Dates: First submitted 2023-10-27; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Neuro-Ophthalmology
Keywords: Virtual reality; Visual field; Ocular alignment; Afferent pupillary function; Efferent pupillary function; Smooth pursuit; Saccades; Gaze holding; Fusional amplitude; Normative data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Healthy volunteers, meaning no known ophthalmological, neurological or vestibular disease.
  The healthy volunteers are within the age groups: 3-6, 7-9, 10-12, 13-17, 18-29, 30-39, 40-49, 50-59, 60-69, 70-79, >80.
- Neurological and ophthalmic patients: Patients with ophthalmological diseases (e.g. strabismus, cataract, macular degeneration, central artery syndrome) Patients with neurological diseases (e.g. Small-Vessel White-Matter Disease, cerebellar ataxia, stroke, downbeat-nystagmus, vascular dementia, multiple sclerosis, M. Parkinson, M. Niemann-Pick type C, M. Alzheimer, galactosemia, schizophrenia, etc).

SUMMARY:
The goal of this clinical study is to collect standard data for the medical device neos™.

neos™ is a system that shows images and measures the resulting eye movements and pupil size.

Collecting standard data involves three steps. First it is checked if neos™ eye-tracking works well. Eye-tracking means recording where a person is looking. After that it is checked if participants look at the images shown in neos™ as planned. Finally the eye movements and the pupil size are measured. This is done in healthy volunteers including children and persons with eye and brain problems.

Participants in the study will wear a virtual reality headset. The screens in the headset will show different images. Cameras in the headset will record eye movements and pupil size. This will take about 15 minutes. During these 15 minutes the investigator looks at the following behaviors of the participants eyes:

* Where are the eyes looking
* How do the pupils react to light and darkness
* How do the eyes move
* How much can the participant see from the corner of their eyes
* How well are the eyes working together

DETAILED DESCRIPTION:
This is a post-market clinical investigation with the overall objective to collect normative data for neos™, including confirming the performance of the neos™ eye-tracking and the adequacy of the neos™visual stimuli.

This clinical investigation also has an exploratory component, looking at the presence of biomarkers in the neos™ examination results.

neos™ is a reusable medical device, that presents visual stimuli to both eyes individually, and measures the resulting eye movements and pupillary changes of each eye.

neos™ is indicated to quantitatively measure:

* The visual field
* Ocular alignment
* Afferent pupillary function
* Efferent pupillary function
* Smooth pursuit (eye movements)
* Saccades (eye movements)
* Gaze holding
* Fusional amplitude

Participants will be recruited within three groups (including children, adolescents and adults):

* Healthy volunteers, meaning no known ophthalmological, neurological or vestibular disease
* Patients with ophthalmological diseases (e.g. strabismus, cataract, macular degeneration, central artery syndrome)
* Patients with neurological diseases (e.g. Small-Vessel White-Matter Disease, cerebellar ataxia, stroke, downbeat-nystagmus, vascular dementia, multiple sclerosis, M. Parkinson, M. Niemann-Pick type C, M. Alzheimer, galactosemia, schizophrenia, etc).

The approximate duration of the single study visit is 25 minutes, not taking the time for patient information and informed consent into account. A follow up period of 15 days exists for the collection of biomarkers recorded in the participant's health record.

The direct clinical benefit from participating in this clinical investigation is the additional information provided by the neos™ examination.

ELIGIBILITY:
Inclusion Criteria Healthy Volunteers:

* Age > 3
* Informed consent by participant and/or legal representative documented per signature
* Snellen visual acuity ≥ +0.1 LogMAR, with correction, on both eyes
* Refractive error between -10 and +5 diopters, on both eyes

Exclusion Criteria Healthy Volunteers:

* Known ophthalmological, neurological or vestibular disease
* Current medication/drugs that could potentially influence performance in ocular motor tasks and/or compliance in the judgement of the investigator (e.g. benzodiazepines, alcohol, or stimulants)
* Stimulative medication (e.g. with Ritalin®)
* Known substance abuse

Inclusion Criteria Patients:

* Age > 3
* Informed consent by participant and/or legal representative, designated trusted person or next of kin, documented per signature
* Refractive error between -10 and +5 diopters, on both eyes
* Known ophthalmological or neurological disease

Exclusion Criteria Patients:

* Visual acuity in one or both eyes < +1.3 LogMAR
* Incapacity to understand and comply with the examination in the opinion of the investigator (e.g. due to very advanced dementia, with failure to comply with easy experimental instructions and tasks)
* Known substance abuse

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The recruitment of healthy volunteers will take place at medical and non-medical sites through advertisement.
  The recruitment of neurological and ophthalmic patients will take place at medical sites through the Principal Investigator.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Normative Datasets | Single study visit - Day 0
  The primery outcome of this post-market clinical investigation is not the testing of a hypothesis, but the collection of normative data for the diagnositic system neos™.
  Normative datasets consisting of Demographic information (age and sex, ethnicity) neos™ output data, i.e. the neos™ report, including the measurement data used to generate the report and data logs generated during the examination.

SECONDARY OUTCOMES:
Accuracy and precision of eye gaze direction | Single study visit - Day 0
  Accuracy and precision of eye gaze direction is calculated from the combination of measurement data and stimuli data applying the methodology described in "Tobii Technology (2011), Accuracy and precision test method for remote eye trackers, Test specification V.2.1.1; February 7th 2011" Will be estimated for the following participant groups
  * Healthy volunteers
  * Patients
  * As a function of interpupillary distance
  * Per age group
Accuracy and precision of pupil size | Single study visit - Day 0
  The accuracy and precision of pupil size is based on the recorded images of the eyes and the independent measurement of the iris diameter.
  Will be estimated for the following participant groups
  * Healthy volunteers
  * Patients
  * As a function of interpupillary distance
  * Per age group
Adequate stimuli | Single study visit - Day 0
  The confirmation of adequate visual stimuli is performed based on the neos™ report. The results presented in the report are assessed against predefined criteria. Adequacy of visual stimuli is reported as a proportion of participants, with 95% confidence interval, for which the adequacy of the visual stimuli was confirmed.
  Will be estimated for the following participant groups:
  * Healthy children (age younger than 13)
  * Healthy adolescents and adults (age older than 13)
  * Per age group
Neuro-ophthalmological biomarkers | Within 30 days before single visit and 14 days after visit
  Neuro-ophthalmological biomarkers present in the participants' medical records are collected. This is an exploratory outcome and will be reported in a frequency table.
neos™ biomarkers | Within 14 days after single visit
  The following biomarkers are expected to be identifiable in the neos™ report:
  Examination block 1: Gaze directions Gaze holding Ocular alignment
  Examination block 2: Pupillary function Efferent pupillary function Afferent pupillary function
  Examination block 3: Eye movements Saccades Smooth pursuit
  Examination block 4: Visual field
  Examination block 5: Fusional amplitude
Comparison of observed and expected biomarkers in ophthalmological and neurological Diseases | Within 14 days after single visit
  For a set of pre-defined ophthalmological and neurological diseases, the presence of biomarkers in the neos™ measurements and in the health record is compared to the expected presence or frequency of biomarkers according to a pre-defined list of biomarkers.

OTHER OUTCOMES:
Safety Outcome | Single study visit - Day 0
  Adverse events and adverse device effects, including any serious adverse events or serious adverse device effects.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Bremova-Ertl, MD, PhD, Principal Investigator — Inselspital
Locations (3):
- Switzerland (3):
  - machineMD AG, Bern, Canton of Bern
  - Inselspital, Bern university hospital, Bern, Canton of Bern
  - Onovis Augenpraxis, Bern, Canton of Bern

REFERENCES:
- See also: Declaration of Helsinki, Version October 2013; — https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- See also: EN ISO 14155: Clinical investigation of medical devices for human participants - Good clinica00l practice, EN ISO 10993: Biological evaluation of medical devices, EN ISO 14971: Application of risk management to medical devices — https://www.iso.org/home.html
- See also: Medical Device Regulation (EU) 2017/745 — https://eur-lex.europa.eu/legal-content/EN/TXT/?uri=CELEX%3A32017R0745
- See also: Tobii Technology (2011), Accuracy and precision test method for remote eye trackers, Test specification V.2.1.1; February 7th 2011 — https://stemedhub.org/resources/3311/download/Tobii_Test_Specifications_Accuracy_and_Pr